CLINICAL TRIAL: NCT00984464
Title: A Phase 2 Study of Intravenous Administration of REOLYSIN (Reovirus Type 3 Dearing) in Combination With Paclitaxel and Carboplatin in Patients With Metastatic Melanoma
Brief Title: Study of REOLYSIN® in Combination With Paclitaxel and Carboplatin in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 020
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Melanoma
Keywords: metastatic; melanoma; REOLYSIN; chemotherapy; carboplatin; paclitaxel
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — reolysin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN — 3x10E10 TCID50, 1 hour intravenous infusion, administered on Days 1,2,3,4 and 5 of a 21-day cycle
Drug: Carboplatin — 6 AUC mg/ml min, 30-min intravenous infusion, given on Day 1 of a 21-day cycle
  Other Names: Paraplatin®
Drug: Paclitaxel — 200 mg/m2, 3-hour intravenous infusion, given on Day 1 of a 21-day cycle
  Other Names: Taxol®

SUMMARY:
The purpose of this Phase 2 study is to investigate whether intravenous administration of REOLYSIN therapeutic virus in combination with paclitaxel and carboplatin is effective and safe in the treatment of metastatic melanoma.

DETAILED DESCRIPTION:
Cutaneous melanoma is one of the most rapidly increasing cancers in the US and around the world with an increase in incidence of about 3-7% per year for fair-skinned Caucasian populations. An estimated 62,480 cases of invasive melanoma will be diagnosed in the US in 2008 with an estimated 8,420 deaths. An additional 46,170 cases of melanoma in situ are predicted.

Melanoma that has spread to distant sites (stage IV) is rarely curable.

This Phase 2 study is designed to characterize the efficacy and safety of REOLYSIN given intravenously in combination with paclitaxel and carboplatin every 3 weeks in patients with metastatic melanoma.

Response is a primary endpoint of this trial.

Patients may continue to receive chemotherapy in combination with REOLYSIN for up to 8 cycles and may continue indefinitely on REOLYSIN monotherapy under this protocol, provided they have not experienced either progressive disease or unacceptable drug-related toxicity that does not respond to either supportive care or dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* have histologically or cytologically confirmed metastatic malignant melanoma.
* have measurable disease.
* have failed at least one prior treatment for metastatic disease or not considered a candidate for standard first line treatment.
* have not received previous carboplatin and/or paclitaxel chemotherapy.
* have NO continuing acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures.
* any surgery involving the melanoma (except biopsies) must have occurred at least 28 days prior to study enrolment.
* be at least 18 years of age.
* have received NO chemotherapy, radiotherapy, immunotherapy or hormonal therapy within 28 days prior to receiving study drug
* have ECOG Performance Score of ≤ 2.
* have a life expectancy of at least 3 months.
* absolute neutrophil ≥ 1.5 x 10^9; Platelets ≥ 100 x10^9; Hemoglobin ≥ 9.0 g/dL; Serum creatinine ≤ 1.5 x upper limit of normal (ULN); Bilirubin ≤ 1.5 x ULN; AST/ALT ≤ 2.5 x ULN.
* negative pregnancy test for females with childbearing potential.
* be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria:

* receive concurrent therapy with any other investigational anticancer agent while on study.
* be good candidate for surgery with curative intent for metastatic disease.
* have a history of or current evidence of brain metastasis(es).
* be on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* be a pregnant or breast-feeding woman.
* have clinically significant cardiac disease.
* have dementia or altered mental status that would prohibit informed consent.
* have any other acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Determine the antitumor effect in terms of objective response rates (i.e., partial response (PR) and complete response (CR) to treatment) | must be confirmed 4 weeks after the criteria for response are first met.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the treatment regimen in the study population. | Within 30 days of last dose of REOLYSIN
Assess progression-free survival (PFS) and overall survival (OS) and disease control [CR+PR+Stable Disease (SD)] rate and duration in the study population | until death

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, MD, PhD, Principal Investigator — Cancer Therapy & Research Center at UTHSCSA
Locations (1):
- Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas, United States